CLINICAL TRIAL: NCT05592314
Title: Lnfluence of the Prosthetic Emergence Profile on the Prevalence of Peri-implant Diseases: a Cross Sectional Study
Brief Title: Lnfluence of the Prosthetic Emergence Profile on the Prevalence of Peri-implant Diseases
Status: Recruiting | Type: Observational
Sponsor: Ramón Pons Calabuig (Other)
Responsible Party: Sponsor-Investigator, Ramón Pons Calabuig, Clinica Professor, Universitat Internacional de Catalunya
Organization: Universitat Internacional de Catalunya (Other)
Other Study IDs: PER-ECL-2020-09a
Record Dates: First submitted 2022-10-19; First posted 2022-10-24 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Peri-Implantitis
Keywords: Dental Implant; Dental prosthesis; Implant-supported; Prevalence; Risk factors
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: No intervention — No intervention

SUMMARY:
1. Objectives:

   To evaluate the influence of the shape and contour of implant-supported restorations on peri-implant soft and hard tissues by using an intraoral scanner.
2. Material and methods:

   1. Number of patients to be treated: 120
   2. Number of visits per patient: 1
   3. Brief description of the different techniques used in the study, authorized and validated in the literature (3-5 lines).

      A clinical and radiographic evaluation of the dental implants of those patients who are undergoing maintenance therapy treated by the Department of Periodontics of the International University of Catalonia prior to 2017 will be carried out. Additionally, a digital scan of the crown will be carried out using a intraoral scanner. Finally, patients will fill out a questionnaire about their routine dental care.
   4. Benefits and harms of participating in the study for the patient

      Participating in this study implies irradiating the patient through a periapical x-ray in order to assess the bone level of their implants and therefore be able to diagnose the presence or absence of peri-implant disease. Regarding the possible benefits, the patient will help the scientific community to determine the ideal contour and shape of the implant-supported restoration that will prevent the appearance of peri-implant diseases. Likewise, patients will undergo an exhaustive clinical and radiographic review that will allow their dental and periodontal status to be updated.
   5. Alternative treatment in case the patient does not wish to participate in the clinical study

      As this is an observational study, there is no alternative treatment. The patient will have absolute freedom to decline to participate in the study.
   6. Treatment to be carried out in the event that complications arise in the patient, once the clinical study has begun

      If after handling the prosthesis, it is detected that any of the screws that support the prostheses are loose or defective, the MORE department will be informed in order to replace said accessory. On the other hand, they would be informed in the same way in case of detecting any complication/alteration with the patient's implant-supported crowns.
   7. Material needed to carry out the study (

   To carry out this study, you will need posterior radiographic positioners, radiographs, an intraoral scanner (3Shape Trios®), the implant analogs or replicas, and a basic periodontal examination set (exploratory probe, periodontal probe, Nabers probe, mirror). and tweezers).
3. Evaluation of experimental and statistical results (3 lines) -

The data obtained will be analyzed through a descriptive statistical analysis (mean, median and standard deviations). The qualitative variables will be expressed in frequencies and percentages. In addition, logistic regression analyzes will be performed to determine the association between peri-implant status (at the implant and patient level) and the angle/emergence of implant-supported prostheses.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18-80 years,
* Implant properly positioned (≥ 2 mm from the buccal plate and >1 mm from the lingual plate or in the ideal occlusal plane horizontally, 5 to 2 mm from the adjacent CEJ or from 2 mm below the residual ridge to crestal position (0 mm) apico-coronally and with an angulation of 70 to 90 degrees from the adjacent tooth long axis or from the ridge parallelism) (21),
* Implant loading for more than 3 years,
* Partial or total edentulism being restored with dental implants in the molar and premolar region with single or partial restorations.
* Patients who have not taken any antibiotic and regular NSAIDs in the last 2 months prior to the clinical examination,

Exclusion Criteria:

* Uncontrolled systemic diseases (i.e., diabetes mellitus)
* Pregnancy or lactation patients,
* Smokers of ≥10 cig/day.
* Zygomatic or pterygoid implants,
* Removable prostheses and cement-retained implant prostheses,
* Patients who have undergone non-surgical peri-implant treatment with prosthesis modifications, peri-implantitis surgical treatment or soft tissue augmentation procedures at the implant site.
* Intake of medications known to modify bone metabolism (i.e., hyperparathyroidism, osteoporosis, and vitamin D deficiency),
* Uncontrolled or active periodontal disease that required treatment.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: patient presents at least one implant-supported restoration in the posterior region (molars and premolars), placed at the university between 2010 and 2017.
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2021-05-05 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Evaluate the influence of excessively contour or overcontoured restorations | February 2021 - may 2023
  Defined as those that present an emergency profile with a marked emergency angle and/or convex profile evaluated by intraoral scanning, in the risk of suffering from peri-implant diseases

CONTACTS AND LOCATIONS:
Locations (1):
- Universitat Internacional de Catalunya, Sant Cugat del Vallès, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: Yes